CLINICAL TRIAL: NCT02065921
Title: Swiss Chronic Obstructive Pulmonary Disease (COPD) Management Cohort COPD-Management: Eine Klinisch-epidemiologische Verlaufsbeobachtung in Hausarztpraxen
Brief Title: Swiss Chronic Obstructive Pulmonary Disease (COPD) Management Cohort
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Prof. Dr. Jörg Leuppi (Other)
Responsible Party: Sponsor-Investigator, Prof. Dr. Jörg Leuppi, Chief of University medical Department Cantonal Hospital Baselland, Cantonal Hosptal, Baselland
Organization: Cantonal Hosptal, Baselland (Other)
Other Study IDs: EKBB170/06
Record Dates: First submitted 2014-02-14; First posted 2014-02-19 (Estimated); Last update posted 2023-09-06 (Actual); Status verified 2023-09

CONDITIONS: Chronic Obstructive Pulmonary Disease; COPD Exacerbation
Keywords: COPD cohort; COPD management; exacerbation
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- COPD patients: establishing COPD cohort database to allow high quality research on diagnosis, treatment, complication and progression of COPD on long-term course.

SUMMARY:
1. Background Chronic Obstructive Pulmonary Disease (COPD) is an inflammatory disease of the lungs, which is most commonly caused by smoking. It is characterized as not fully reversible airflow limitation, chronic cough and dyspnoea. Being the fourth leading cause of death worldwide, COPD is an important public health challenge and can be prevented and treated. It is estimated that at least 400,000 individuals in Switzerland are affected by COPD. This number may increase in the coming years due to increasing nicotine consumption.

   In response to the rising trend, the Global Initiative for Chronic Obstructive Lung Disease (GOLD) has established new guidelines on the global strategy for diagnosis, management and prevention of COPD. Systematic diagnosis and stratification are crucial for effective treatment measures.

   As COPD is an irreversible and progressive disease, its treatment aims an early detection and better management, which leads preventing progression. Disease management programs have shown that only patients who understand their exacerbation symptoms can benefit. Moreover, it is a major goal to improve health-related quality of life by reducing symptoms and decelerating disease progression.

   Spirometry is the golden standard for the diagnosis of COPD, to assess the severity of the obstruction, and as a guide for optimal therapeutic measures.
2. Aim of the study The objective of this project is to establish a COPD cohort database to allow high quality research on diagnosis, treatment, complication and progression of COPD on long-term course.

   Spirometry should be used consistently for the diagnosis and the monitoring of the development of the disease. Using collected information such as spirometric data, disease progression's data and therapeutic measures should help improve the management and self-management of the patients.
3. Methods 3.1 Study design We are conducting a prospective cohort study, based on COPD patients from northern and western Switzerland, who are managed under primary care setting. Patients with mild to very severe COPD (GLOD stages I-IV) are enrolled in the study.

   Currently, 67 General practitioners (GPs) are participating in our Study. Each GP recruits 1-20 patients with presumed mild to very severe COPD according to criteria of the Global Initiative for Chronic Obstructive Lung disease [GOLD].

   Patients' follow-up-visits occurs at 6-month intervals; their history, symptoms and examination status is recorded. Data is entered into an online database either by the physicians or by study team after receiving the collected data questionnaires by facsimile.

   Data collection includes demographic data, physical examination, spirometric parameters, medical treatment and exacerbation history besides death.

   A spirometer (EasyOne™, ndd Medizintechnik AG, Zürich, Switzerland) is used to assess lung function. All participating physicians were instructed on the usage of the spirometer and on how to complete spirometry according to the guidelines. For the assessment of the severity of COPD, we use the spirometric data provided by the GPs. The COPD severity is interpreted according to criteria of the GOLD committee.

   3.2 Patient population Patients with newly diagnosed or existing COPD, who are managed in primary-care practices.

   3.3 Inclusion criteria
   * Tiffenau (FEV17FVC) < 70 without reversibility (Increase in FEV1 after inhalation of a bronchodilator <200 ml and <12%).
   * Age: > 40 years
   * Both genders
   * Smokers or ex-smokers of at least 20 pack years.
   * Informed consent.

   3.4 Archiving and Data Retention All study-related records such as medical records, informed consent documents, information regarding participants who discontinued, and other pertinent data will be maintained and therefore retained as long as required by the applicable Swiss regulatory requirements (10 Years).

   3.5 Data security The complete data of the study will be entered anonymously into a database. The data is password-protected and can only be accessed by investigators and study members.
4. Publication and authorship 4.1 Publication policy

Authorship credit is based on:

1. Substantial contribution to conception and design, acquisition of data, or analysis and interpretation of data.
2. Drafting the article or revising it critically for important intellectual content.
3. Final approval of the version to be published. Each author should have participated sufficiently in the work to take public responsibility for appropriate portions of the content.

ELIGIBILITY:
Inclusion Criteria:

* Tiffenau (FEV17FVC) < 70 without reversibility (Increase in FEV1 after inhalation of a bronchodilator <200 ml and <12%).
* Age: > 40 years
* Both genders
* Smokers or ex-smokers of at least 20 pack years.
* Informed consent.

Exclusion Criteria:

* < 40 Years
* Tiffenau (FEV17FVC) > 70

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with newly diagnosed or existing COPD, who are managed in primary-care practices.
Sampling Method: Non-Probability Sample
Enrollment: 265 (Estimated)
Dates: Start 2006-09; Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Number of exacerbation | 24 months
  no. of exacerbation and time to exacerbation over a time period of 2 years.

SECONDARY OUTCOMES:
Disease progression | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Cantonal Hospital Baselland, Internal medicine University clinic, Liestal, Basel-Landschaft, Switzerland

REFERENCES:
- [Result] Jochmann A, Scherr A, Jochmann DC, Miedinger D, Torok SS, Chhajed PN, Tamm M, Leuppi JD. Impact of adherence to the GOLD guidelines on symptom prevalence, lung function decline and exacerbation rate in the Swiss COPD cohort. Swiss Med Wkly. 2012 Apr 5;142:w13567. doi: 10.4414/smw.2012.13567. eCollection 2012. PMID 22481636
- [Result] Jochmann A, Neubauer F, Miedinger D, Schafroth S, Tamm M, Leuppi JD. General practitioner's adherence to the COPD GOLD guidelines: baseline data of the Swiss COPD Cohort Study. Swiss Med Wkly. 2010 Aug 9;140:10.4414/smw.2010.13053. doi: 10.4414/smw.2010.13053. eCollection 2010. PMID 20407960
- [Derived] Urwyler P, Abu Hussein N, Bridevaux PO, Chhajed PN, Geiser T, Grendelmeier P, Joos Zellweger L, Kohler M, Maier S, Miedinger D, Tamm M, Thurnheer R, Dieterle T, Leuppi JD. Predictive factors for exacerbation and re-exacerbation in chronic obstructive pulmonary disease: an extension of the Cox model to analyze data from the Swiss COPD cohort. Multidiscip Respir Med. 2019 Feb 5;14:7. doi: 10.1186/s40248-019-0168-5. eCollection 2019. PMID 30774953